CLINICAL TRIAL: NCT07223281
Title: Real-World Effectiveness of Amniotic Membrane Allografts Versus Standard Wound Care in Chronic Wound Healing: A Multi-Site Study in Diabetic Foot Ulcers (DFU), Venous Leg Ulcers (VLU), and Pressure Ulcers (PU)
Brief Title: Real-World Effectiveness of Amniotic Membrane Allografts Versus Standard Wound Care in DFU, VLU, and PU
Status: Active, not recruiting | Type: Observational
Sponsor: Legacy Medical Consultants (Industry)
Responsible Party: Sponsor
Other Study IDs: LMCRWE25
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Venous Leg Ulcers (VLUs); Pressure Ulcers, Bedsores, Decubitus Ulcer
Keywords: real world evidence; wound healing
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- Zenith™ + Standard care for DFU: Patients who received Zenith™ plus standard care for their DFU
- Orion™ + Standard care for DFU: Patients who received Orion™ plus standard care for their DFU
- SurGraft FT™ + Standard care for DFU: Patients who received SurGraft FT™ plus standard care for their DFU
- Complete ACA™ + Standard care for DFU: Patients who received Complete ACA™ plus standard care for their DFU
- Standard care alone for DFU: Patients who received standard care only for their DFU
- Zenith™ + Standard care for VLU: Patients who received Zenith™ plus standard care for their VLU
- Orion™ + Standard care for VLU: Patients who received Orion™ plus standard care for their VLU
- SurGraft FT™ + Standard care for VLU: Patients who received SurGraft FT™ plus standard care for their VLU
- Complete ACA™ + Standard care for VLU: Patients who received Complete ACA™ plus standard care for their VLU
- Standard care alone for VLU: Patients who received standard care only for their VLU
- Zenith™ + Standard care for PU: Patients who received Zenith™ plus standard care for their PU
- Orion™ + Standard care for PU: Patients who received Orion™ plus standard care for their PU
- SurGraft FT™ + Standard care for PU: Patients who received SurGraft FT™ plus standard care for their PU
- Complete ACA™ + Standard care for PU: Patients who received Complete ACA™ plus standard care for their PU
- Standard care alone for PU: Patients who received standard care only for their PU

SUMMARY:
This observational study will evaluate the real-world effectiveness of four amniotic membrane-based products (Zenith™, Orion™, SurGraft FT™, Complete ACA™) in addition to standard care, compared with standard care alone. The study will use complete electronic health records (EHR) from multiple wound care centers across the United States (2022-2025) to generate study data for product-treated and propensity score-matched standard care cohorts for each product-indication combination. The overall study comprises 12 parallel sub-studies (one for each product-wound type combination), each aiming to answer whether adding the product improves healing outcomes versus standard care alone in that indication. The primary endpoint is the proportion of wounds achieving complete closure within 12 weeks, with subgroup analyses by wound severity measures, age groups, and number of product applications. Secondary outcomes are time-to-healing, early wound improvement (≥50% reduction in wound area by 4 weeks), wound-related complications, and subgroup analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18; DFU/VLU/PU; sufficient observable timeline

Exclusion Criteria:

* Use of other advanced wound products, atypical ulcer etiology (e.g., malignancy, vasculitis); insufficient follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DFU, VLU, or PU
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure at 12 Weeks | From index visit to 12 weeks post-index
  Proportion of index wounds with 100% epithelialization, no drainage or dressings; confirmation on ≥1 follow-up within 60 days

SECONDARY OUTCOMES:
Time to complete wound closure | From index visit up to 24 months post-index
  Time from the index visit to primary complete wound closure for wounds that heal during the study period
≥50% wound area reduction at 4 weeks | From index visit to 4 weeks post-index
  Proportion of patients whose wounds close greater than 50% within 4 weeks from the index visit
Wound-related complications | From index visit up to 24 months post-index
  Wound-related complications including infection requiring treatment, hospitalization, ED visits, and major or minor amputation

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Colorado Foot and Ankle, Colorado Springs, Colorado
  - Podiatric Surgical Specialists, Clinton Township, Michigan
  - Advanced Wound Therapy, Tulsa, Oklahoma
  - Comprehensive Occupational Medicine, Nitro, West Virginia

REFERENCES:
- [Result] Kahoun, J., Gorenstein, S., & Gillette, B. (2025). Real-World Performance of Amniotic Membrane Allografts for Chronic Wounds: Multi-Site Results from a Retrospective EHR Study. https://doi.org/10.5281/zenodo.17504472